CLINICAL TRIAL: NCT06540027
Title: The Effect of Minimally Invasive Surgery on Systemic Inflammatory Response in Rectal Cancer
Status: Enrolling by invitation | Type: Observational
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: basaksehir2024-37
Record Dates: First submitted 2024-08-02; First posted 2024-08-06 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-07

CONDITIONS: Colorectal Cancer; Colorectal Adenocarcinoma; Rectal Cancer; Rectal Cancer Stage; Immune System Disorder
Keywords: minimally invasive surgery; robotic surgery; colorectal cancer; immune system response
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms; Immune System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group: Patients with rectal cancer, open surgery
  Interventions: Procedure: rectal cacer surgery
- Study group 1: Patients with rectal cancer, laparoscopic surgery
  Interventions: Procedure: rectal cacer surgery
- Study group 2: Patients with rectal cancer, robotic surgery
  Interventions: Procedure: rectal cacer surgery

INTERVENTIONS:
Procedure: rectal cacer surgery — minimally invasive surgery

SUMMARY:
As a hypothesis and shown in many meta-analyses and randomized controlled studies, minimally invasive surgery causes less surgical trauma and therefore less proinflammatory response and immunosuppression develop, and postoperative recovery is faster. Although various prognostic studies on the relationship between gastrointestinal cancer types and SII (systemic inflammatory index) and the use of minimally invasive surgery have been published, the high level of this response and the type of surgery in the treatment of colorectal cancer have not yet been shown to have a direct effect on SII.

DETAILED DESCRIPTION:
Minimally invasive surgery has been demonstrated to significantly enhance the host immune response in colorectal cancer. The effect and the SII marker may be reliable indicators of this enhancement. A retrospective analysis was conducted on the records of patients who underwent surgery for colorectal cancer at our clinic over a four-year period. The patients were divided into three groups according to the surgical approach employed: open surgery, laparoscopic surgery and robotic surgery.

The primary outcome is: A comparison of the open surgery group with those undergoing minimally invasive surgery (laparoscopic and robotic) revealed lower SII values in the robotic surgery group than in the laparoscopic surgery group.

The secondary outcome : The SII values were determined as neutrophil/lymphocyte and platelet/lymphocyte, which had been previously investigated in other studies.

A comparison will be made with the relevant markers. The research team adheres to the principles set forth in the Declaration of Helsinki and Good Clinical Practice guidelines. They will conduct the study in an appropriate manner.

No intervention will be made in the follow-up and treatment of patients, in accordance with the approval of the hospital ethics committee.

The laboratory records typically examined in the postoperative phase will be re-examined in a retrospective manner. Furthermore, the personal data of the participants will not be incorporated into the study.

ELIGIBILITY:
Inclusion Criteria:

Patients operated for rectal cancer

* Open surgery
* Laparoscopic surgery
* Robotic surgery

Exclusion Criteria:

* Patients with diagnosed immune deficiency
* Patients with recurrent colorectal cancer
* Patients with co-existent tumors

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients operated with minimally invasive surgery
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
immune response | 1 day
  the level of SII

CONTACTS AND LOCATIONS:
Overall Officials: Serkan Sari, Prof, Study Chair — Basaksehir Cith Hospital, Istanbul, Turkey
Locations (1):
- Yigit Duzkoylu, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: reference — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC9419130/
- See also: reference — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9446812/
- See also: reference — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC8629478/
- See also: reference — http://www.cirugiaycirujanos.com/frame_esp.php?id=666